CLINICAL TRIAL: NCT00384774
Title: A Placebo-Controlled, Group Sequential, Adaptive Treatment Assignment Study of Intravenous COL-144 (LY573144) in the Acute Treatment of Migraine
Brief Title: A Placebo-Controlled Adaptive Treatment Assignment Study of Intravenous COL-144 in the Acute Treatment of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16891; 2006-003903-38 (EudraCT Number); COL MIG-201 (Other: Colucid); H8H-CD-LAHM (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-01

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lasmiditan (Experimental): Participants received escalating doses of 2.5 mg, 5 mg, 10 mg, 20 mg, 30 mg and 45 mg of lasmiditan as intravenous injection.
  Interventions: Drug: Lasmiditan
- Placebo (Placebo Comparator): Participants received intravenous infusion of placebo solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lasmiditan — Administered as intravenous infusion
  Other Names: LY573144, COL-144
  Arms: Lasmiditan
Drug: Placebo — Administered as intravenous infusion
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of a range of intravenous doses of COL-144 in the treatment of migraine headache in order to select a dose range for further studies.

DETAILED DESCRIPTION:
This study is set up:

* to evaluate the efficacy (headache response at two hours) of a range of intravenous doses of COL-144 in order to select a dose range for further evaluation,
* to explore the time course and effect of a range of dose levels of COL-144 on features of the migraine including: headache response, proportion of participants pain-free, headache recurrence, nausea, photophobia, phonophobia, disability, use of rescue medication, patient global impression and vomiting
* to explore the safety and tolerability of a range of doses of COL-144 in terms of adverse events, physical exam, vital signs, laboratory evaluations, and ECGs
* to determine key PK parameters for COL-144 and to explore the relationship between the PK of COL-144 and the time course and extent of clinical response

ELIGIBILITY:
Inclusion Criteria:

* Patients with migraine with or without aura fulfilling the IHS diagnostic criteria 1.1 and 1.2.1 (2004)
* History of migraine of at least 1 year
* Migraine onset before the age of 50 years
* History of 1 - 8 migraine attacks per month
* Male or female subjects aged 18 to 65 years
* Female patients of child-bearing potential must be using a highly effective form of contraception (eg combined oral contraceptive, IUD, abstinence, vasectomized partner)
* Able and willing to return to the clinic for treatment within 4 hours of the onset of a migraine headache
* Able and willing to give written informed consent

Exclusion Criteria:

* History of life threatening or intolerable adverse reaction to any triptan
* Use of prescription migraine prophylactic drugs
* Pregnant or breast-feeding women
* Women of child-bearing potential not using highly effective contraception
* History or evidence of coronary artery disease, ischemic or hemorrhagic stroke, epilepsy or any other condition placing the patient at increased risk of seizures
* History of hypertension (controlled or uncontrolled)
* Sitting BP >160mmHg systolic or >90mmHg diastolic on 2 repeated measurements at screening
* Current use of hemodynamically active cardiovascular drugs
* History within the previous 3 years or current evidence of abuse of any drug, prescription or illicit, or alcohol
* Significant renal impairment
* Previous participation in this clinical trial
* Participation in any clinical trial of an experimental drug or device in the previous 30 days
* Any medical condition or laboratory test which in the judgment of the investigator makes the patient unsuitable for the study
* Relatives of, or staff directly reporting to, the investigator
* Patients with known hypersensitivity to COL-144, other 5HT1F receptor agonists or to any excipient of COL-144

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Helsinki, Finland
- Essen, Germany
- Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Reuter U, Pilgrim A, Diener HC, Färkkilä M, Ferrari M for the European COL-144 investigators. COL-144: A Selective 5-HT1F Agonist For the Treatment of Migraine Attacks. European Headache & Migraine Trust International Congress 2008, London, England, Poster #PC.11, September 5, 2008.
- [Derived] Blumenfeld A, Tepper SJ, Khanna R, Doty E, Vincent M, Miller SI. Serotonin syndrome in the acute treatment landscape of migraine: the lasmiditan experience. Front Neurol. 2023 Oct 27;14:1291102. doi: 10.3389/fneur.2023.1291102. eCollection 2023. PMID 37965170
- [Derived] Ferrari MD, Farkkila M, Reuter U, Pilgrim A, Davis C, Krauss M, Diener HC; European COL-144 Investigators. Acute treatment of migraine with the selective 5-HT1F receptor agonist lasmiditan--a randomised proof-of-concept trial. Cephalalgia. 2010 Oct;30(10):1170-8. doi: 10.1177/0333102410375512. Epub 2010 Jun 15. PMID 20855362

RESULTS

PARTICIPANT FLOW:
Groups:
- Lasmiditan 2.5 mg: Participants received 2.5 mg of lasmiditan administered as intravenous infusion.
- Lasmiditan 5.0 mg: Participants received 5 mg of lasmiditan administered as intravenous infusion.
- Lasmiditan 10 mg: Participants received 10 mg of lasmiditan administered as intravenous infusion.
- Lasmiditan 20 mg: Participants received 20 mg of lasmiditan administered as intravenous infusion.
- Lasmiditan 30 mg: Participants received 30 mg of lasmiditan administered as intravenous infusion.
- Lasmiditan 45 mg: Participants received 45 mg of lasmiditan administered as intravenous infusion.
Period: Overall Study
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Started | 42 | 4 | 12 | 24 | 28 | 16 | 4
Received at Least 1 Dose of Study Drug | 42 | 4 | 12 | 24 | 28 | 16 | 4
Completed | 42 | 4 | 12 | 24 | 28 | 16 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg | Total
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (13.1) | 46.8 (14.0) | 39.2 (8.8) | 34.5 (10.3) | 38.9 (10.1) | 40.3 (11.2) | 40.8 (11.0) | 39.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 3 | 10 | 21 | 24 | 14 | 3 | 113
  Male | 4 | 1 | 2 | 3 | 4 | 2 | 1 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 42 | 4 | 11 | 20 | 28 | 16 | 4 | 125
  Black | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Latin | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  South-American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Romanian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 3 | 0 | 1 | 3 | 1 | 0 | 1 | 9
  Finland | 10 | 0 | 6 | 4 | 2 | 1 | 1 | 24
  Germany | 29 | 4 | 5 | 17 | 25 | 15 | 2 | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Headache Response at Two Hours After Initiation of Infusion of Study Drug
Description: Headache response is a binary response variable derived from the headache intensities recorded in the participant diary. Headache response is defined as a reduction in headache severity from moderate or severe at baseline to mild or no headache, at two hours after initiation of infusion of study drug.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4
Participants
  No | 23 | 2 | 10 | 11 | 10 | 5 | 1
  Yes | 19 | 2 | 2 | 13 | 18 | 11 | 3
Statistical Analysis 1: Comparison: Placebo vs Lasmiditan 2.5 mg; Headache Response; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan 5.0 mg; Headache Response; Test type: Superiority or Other; p = 0.0991, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan 10 mg; Headache Response; Test type: Superiority or Other; p = 0.4851, Chi-squared
Statistical Analysis 4: Comparison: Placebo vs Lasmiditan 20 mg; Headache Response; Test type: Superiority or Other; p = 0.1178, Chi-squared
Statistical Analysis 5: Comparison: Placebo vs Lasmiditan 30 mg; Headache Response; Test type: Superiority or Other; p = 0.1093, Chi-squared
Statistical Analysis 6: Comparison: Placebo vs Lasmiditan 45 mg; Headache Response; Test type: Superiority or Other; p = 0.3364, Fisher Exact

2. Secondary Outcome: Percentage of Participants With Headache Response 10 to 240 Minutes (Min) Post Dose
Description: Headache response is defined as a reduction in headache severity from moderate or severe at baseline to mild or no headache, at two hours after initiation of infusion of study drug.
Time Frame: 10, 20, 40, 60 90, 120, 180 and 240 minutes post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4
Percentage of participants
  10 min | 11.9 | 0 | 8.3 | 8.3 | 14.3 | 12.5 | 75.0
  20 min | 26.2 | 0 | 16.7 | 25.0 | 39.3 | 50.0 | 75.0
  40 min | 35.7 | 0 | 25.0 | 37.5 | 50.0 | 75.0 | 75.0
  60 min | 33.3 | 50.0 | 25.0 | 50.0 | 53.6 | 75.0 | 50.0
  90 min | 47.6 | 50.0 | 25.0 | 45.8 | 53.6 | 68.8 | 75.0
  120 min | 45.2 | 50.0 | 16.7 | 54.2 | 64.3 | 68.8 | 75.0
  180 min | 33.3 | 50.0 | 25.0 | 54.2 | 60.7 | 68.8 | 75.0
  240 min | 31.0 | 75.0 | 33.3 | 54.2 | 57.1 | 68.8 | 25.0

3. Secondary Outcome: Percentage of Participants Headache Free
Description: Headache free is defined as a reduction in headache severity from moderate or severe at baseline to no headache pain at 10 min, 20 min, 40 min, 60 min, 90 min, 120 min, 180 min, and 240 min after initiation of study drug.
Time Frame: 10, 20, 40, 60 90, 120, 180 and 240 minutes post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 27 | 16 | 3
Percentage of participants
  10 min | 0 | 0 | 0 | 0 | 3.6 | 0 | 25.0
  20 min | 2.4 | 0 | 0 | 8.3 | 3.6 | 0 | 25.0
  40 min | 2.4 | 0 | 0 | 8.3 | 14.3 | 18.8 | 25.0
  60 min | 7.1 | 0 | 0 | 20.8 | 21.4 | 25.0 | 25.0
  90 min | 14.3 | 0 | 0 | 20.8 | 25.0 | 37.5 | 25.0
  120 min | 19.0 | 0 | 0 | 20.8 | 28.6 | 37.5 | 25.0
  180 min | 21.4 | 0 | 0 | 20.8 | 32.1 | 37.5 | 25.0
  240 min | 21.4 | 25.0 | 0 | 20.8 | 28.6 | 31.3 | 25.0

4. Secondary Outcome: Number of Participants With Sustained Headache Response
Description: Sustained headache response at 2 hours is a binary response variable derived from the headache intensities recorded in the participant diary. Sustained headache response was defined as moderate or severe headache pain at baseline which became mild or absent (pain free) at 2 hours after initiation of study drug and which did not recur (became moderate or severe) within 24 hours of initiation of study drug. If rescue medication was taken within 24 hours, this was considered a headache recurrence, even if no headache was reported.
Time Frame: 2 to 24 hours post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4
Participants
  No | 29 | 2 | 11 | 16 | 18 | 7 | 3
  Yes | 13 | 2 | 1 | 8 | 10 | 9 | 1

5. Secondary Outcome: Number of Participants With Sustained Pain Free
Description: Sustained pain free was defined as moderate or severe headache pain at baseline which became mild or absent (pain free) at 2 hours after initiation of study drug and which did not recur (became moderate or severe) within 24 hours of initiation of study drug. If rescue medication was taken within 24 hours, this was considered a headache recurrence, even if no headache was reported.
Time Frame: 2 to 24 hours post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4
Participants
  No | 35 | 4 | 12 | 21 | 23 | 13 | 3
  Yes | 7 | 0 | 0 | 3 | 5 | 3 | 1

6. Secondary Outcome: Number of Participants With Absence of Nausea, Vomiting, Photophobia and Phonophobia
Description: Number of participants with absence of nausea, vomiting, photophobia and phonophobia.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4
Participants
  Nausea | 7 | 1 | 5 | 3 | 6 | 1 | 1
  Vomiting | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Photophobia | 21 | 1 | 9 | 11 | 12 | 4 | 1
  Phonophobia | 18 | 1 | 5 | 6 | 7 | 4 | 1

7. Secondary Outcome: Number of Participants With Clinical Disability
Description: Clinical disability for each participant was assessed using the Clinical Disability Questionnaire (CDQ). Participants graded their disability on the following scale: 0, no disability, able to function normally; 1, performance of daily activities mildly impaired, can still do everything but with difficulty; 2, performance of daily activities moderately impaired, unable to do some things; 3, performance of daily activities severely impaired, cannot do all or most things, bed rest may be necessary.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4
Participants
  No disability | 11 | 2 | 1 | 6 | 9 | 7 | 3
  Mild disability | 10 | 1 | 1 | 7 | 7 | 5 | 0
  Moderate disability | 14 | 0 | 6 | 7 | 11 | 3 | 0
  Severe disability | 7 | 1 | 4 | 4 | 1 | 1 | 1

8. Secondary Outcome: Percentage of Participants Using Rescue Medication
Description: Use of rescue medication up to 24 hours after initiation of study drug.
Time Frame: 24 hours post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4
Percentage of participants | 69.0 | 25.0 | 91.7 | 58.3 | 53.6 | 37.5 | 25.0

9. Secondary Outcome: Percentage of Participants Reporting a Score on the Patient Global Impression (PGI)
Description: PGI scale is a participant-rated instrument that measures participants own global impression of their illness severity. Participants were asked to mark the box that best describes their headache condition since they started taking the medicine. The options in the displayed boxes are represented on a 7-point scale, with 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
Number analyzed (Participants) | 42 | 4 | 12 | 24 | 28 | 16 | 4
Percentage of Participants
  Very much better | 9.5 | 0 | 0 | 8.3 | 25.0 | 37.5 | 0
  Much better | 19.0 | 75.0 | 8.3 | 29.2 | 17.9 | 31.3 | 50.0
  A little better | 23.8 | 0 | 41.7 | 29.2 | 42.9 | 18.8 | 25.0
  No change | 19.0 | 0 | 25.0 | 29.2 | 7.1 | 12.5 | 25.0
  A little worse | 14.3 | 0 | 8.3 | 4.2 | 7.1 | 0 | 0
  Much worse | 11.9 | 0 | 0 | 0 | 0 | 0 | 0
  Very much worse | 2.4 | 25.0 | 16.7 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up To 7 Days
Description: All randomized participants who received at least one dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- Placebo: Participants received intravenous injection of placebo solution.
Arm/Group | Placebo | Lasmiditan 2.5 mg | Lasmiditan 5.0 mg | Lasmiditan 10 mg | Lasmiditan 20 mg | Lasmiditan 30 mg | Lasmiditan 45 mg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/4 | 0/12 | 0/24 | 0/28 | 0/16 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/4 | 0/12 | 0/24 | 0/28 | 0/16 | 0/4
Other Adverse Events (participants affected / at risk) | 18/42 | 2/4 | 3/12 | 17/24 | 19/28 | 13/16 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=42) | Lasmiditan 2.5 mg (N=4) | Lasmiditan 5.0 mg (N=12) | Lasmiditan 10 mg (N=24) | Lasmiditan 20 mg (N=28) | Lasmiditan 30 mg (N=16) | Lasmiditan 45 mg (N=4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 3 (3) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 3 (3) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling of relaxation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Infusion site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensation of blood flow (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2) | 1 (1) | 8 (9) | 7 (7) | 3 (4) | 1 (1)
Formication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 8 (11) | 3 (4) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phonophobia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 1/38 (1) | 0/3 (0) | 0/10 (0) | 0/21 (0) | 0/24 (0) | 0/14 (0) | 0/3 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasoconstriction (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the Study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.